CLINICAL TRIAL: NCT06680050
Title: AUSTRAL Trial: An Open-Label, Multicenter, Phase II Study Of Radiotherapy Followed By Durvalumab (MEDI4736) And Ceralasertib (AZD6738) In Stage III NSCLC Patients With Thoracic Relapses +/- Oligometastases After PACIFIC Regimen
Brief Title: Phase II Study of Radiotherapy Followed by Durvalumab and Ceralasertib in Stage III NSCLC Patients With Thoracic Relapses +/- Oligometastases After PACIFIC Regimen
Acronym: AUSTRAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-515942-18-01
Record Dates: First submitted 2024-10-30; First posted 2024-11-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer NSCLC
MeSH Terms: interventions — durvalumab; ceralasertib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiotherapy followed by Durvalumab+Ceralasertib (Experimental)
  Interventions: Drug: Durvalumab (MEDI4736); Drug: Ceralasertib; Radiation: radiotherapy

INTERVENTIONS:
Drug: Durvalumab (MEDI4736) — Durvalumab will be administered via IV infusion at a dose of 1500 mg on day 8 Q4W until confirmed disease progression unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.
Drug: Ceralasertib — Ceralasertib dose will be administered orally, 240mg BID, approximately 12 ± 2 hours apart, days 1 to 7 q28 (Q4W), up to progression or unacceptable toxicity.
Radiation: radiotherapy — Loco-regional recurrences of the primary tumor and regional lymph node metastases will be treated with a total dose of 36 to 50 Gy in daily fractions with a dose of 2 to 3 Gy per fraction. Two weeks from the last dose of radiotherapy, a systemic treatment with durvalumab and ceralasertib will be started.

SUMMARY:
Aim of this phase 2 study is to explore the safety and efficacy of thoracic re-irradiation +/- SBRT to oligometastases (<3) followed after an interval of 2 weeks by durvalumab and ceralasertib for patients with thoracic relapses +/- oligometastases after PACIFIC or PACIFIC-like (concurrent or sequential chemo-radiotherapy followed by maintenance durvalumab) regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed, written and dated informed consent and any locally required authorization
2. Male or female aged 18 years or older
3. ECOG Performance Status of 0-2
4. Life expectancy ≥ 6 months at the start of treatment
5. Body weight >30kg
6. Maintenance treatment with durvalumab for a minimum of 3 months
7. Histologically or cytologically documented locally advanced NSCLC at relapse
8. Measurable disease as defined by RECIST v1.1
9. Documented tumor cell PD-L1 status at first diagnosis and/or at relapse
10. Thoracic progression as defined by PACIFIC protocol, with or without a maximum of 3 metastatic lesions amenable to local radiotherapy (at discretion of treating center)
11. Interval of > 12 months between the end of the first thoracic radiotherapy (PACIFIC)
12. Pre-treatment whole body CT scan with i.v. contrast medium
13. Pre-treatment CT-PET scan
14. Pre-treatment brain MRI
15. Evidence of post-menopausal status, or negative urinary/serum pregnancy test for female pre-menopausal patients
16. Patient willing and able to comply with the protocol procedures for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Patients who discontinued durvalumab due to local or systemic progression during the maintenance phase < 12 months after the end of CRT
2. Patients who experienced, during the maintenance phase with durvalumab after CRT, grade 3 or more documented immune-related toxicity (with the exception of fully recovered endocrine toxicities) or grade 3 or more radiation-induced pneumonitis.
3. Any unresolved toxicity NCI CTCAE from previous anticancer therapy not completely resolved or not resolved to baseline prior to screening for this study with the exception of alopecia, vitiligo, and the laboratory values defined below

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
   3. Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
4. Any toxicity that led to permanent discontinuation of prior immunotherapy
5. Patients with more than 3 distant metastases (non-oligometastatic disease)
6. Patients with metastatic disease progression not amenable for radical radiotherapy such as malignant ascites, pleural or pericardial effusion, diffuse lymphangiosis of skin or lung, diffuse bone marrow metastasis, metastasis invading the GI tract, abdominal masses/abdominal organomegaly, identified by physical exam that is not measurable by reproducible imaging techniques.
7. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
8. Diagnosis of ataxia telangiectasia
9. Patients harboring targetable genomic alterations, such as EGFR, HER-2 or MET exon14 skipping mutations, ALK, ROS1, RET or NTRK rearrangements. Molecular profiling can be assessed on archival tumor samples or on new tissue or liquid biopsy.
10. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
11. Concurrent participation (including the follow-up period) in another clinical study with an investigational product or during the last 4 weeks unless it is an observational (non-interventional) clinical study.
12. Any concurrent chemotherapy, immunotherapy, biological or hormonal therapy only for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
13. Inadequate bone marrow reserve or organ function as defined below:

    1. Absolute neutrophil count <1.5 x 109/L (1500/mm3)
    2. Platelets <100 x 109/L (100000/mm3)
    3. Haemoglobin <9.0 g/dL (5.59 mmol/L)
    4. Serum bilirubin <1.5 x upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinaemia that is predominantly unconjugated in the absence of evidence of haemolysis or hepatic pathology) who will be allowed in consultation with their physician.
    5. AST and ALT <2.5 x ULN.
    6. Inadequate renal function: measured creatinine clearance (CL) <40 ml/min or calculated CL (according to Cockroft-Gault): <40ml/min or by 24-hour urine collection for determination of CL
14. History of active primary immunodeficiency
15. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

1. Patients with vitiligo or alopecia 2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement 3. Any chronic skin condition that does not require systemic therapy 4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician 5. Patients with celiac disease controlled by diet alone 16. Female patients who are pregnant, breast-feeding, male, or female patients of reproductive potential who are not employing an effective method of birth control from screening to 90 days after the last dose of durvalumab.

17. History of allogenic organ transplantation 18. Any condition that, in the opinion of the Investigator, would interfere with the evaluation of the study drug or interpretation of patient safety or study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability, in terms of number of grade 3 or higher adverse events judged as at least possibly related to study treatment regimen | within 6 months from the start of study treatment
PFS | 12 months
  PFS is defined as the time from the date of enrolment until the date of first disease progression or death to any cause, whichever comes first.

SECONDARY OUTCOMES:
ORR | 12 months
  Objective response is defined as either complete response (CR) or partial response (PR) as determined by the investigator
Efficacy in terms of PFS rate | 6 and 12 months
Efficacy in terms of OS | 6 and 12 months
  OS is defined as the time from enrolment until the date of death from any cause
Efficacy in terms of OS rate | 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (7):
  - ASST degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - IRCCS Ospedale Policlinico San Martino, Genova, Genova
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda ospedaliera di Padova, Padua
  - Azienda Ospedaliero - Universitaria di Parma, Parma
- Switzerland (2):
  - University Hospital of Geneva, Geneva
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Filippi AR, Rulli E, Signorelli D, Willmann J, Durham A, De Simone I, Santoni A, Galli F, Carlucci L, Torri V, Lo Russo G, Addeo A, Guckenberger M. Rationale and Design of the AUSTRAL trial: An Open-Label, Multicenter, Phase II Study Evaluating Radiotherapy Followed by Durvalumab (MEDI4736) and Ceralasertib (AZD6738) in Stage III NSCLC Patients With Thoracic Relapses and/or Oligometastases After the PACIFIC Regimen. Clin Lung Cancer. 2025 Dec;26(8):e633-e638. doi: 10.1016/j.cllc.2025.07.006. Epub 2025 Jul 12. PMID 40781023